CLINICAL TRIAL: NCT06454643
Title: The Pharmacological and Clinical Aspects of Using Gentamicin in Cardiac Surgery
Brief Title: Gentamicin in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Rasheed University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AR200311
Record Dates: First submitted 2024-05-26; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Infection
Keywords: infection; antibiotics; antimicrobial prophylaxis; aminoglycoside; Gentamicin
MeSH Terms: conditions — Infections | interventions — Floxacillin; Gentamicins; Ceftriaxone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Patients received flucloxacillin and ceftriaxone 60 minute before incision and then continued for 48 hours as follows:
  * Flucloxacillin 2g given before surgery then 1g * 4 for 48 hours after operation.
  * Ceftriaxone 1g given before surgery then 1g * 2 for 48 hours after operation.
  Interventions: Drug: Flucloxacillin and ceftriaxone
- Gentamicin (Experimental): Patients received flucloxacillin and gentamicin 60 minute before incision and then continued for 48 hours, as follows:
  * Flucloxacillin 2g given before surgery then 1g * 4 for 48 hours after operation.
  * Gentamicin 2mg/kg of ideal body weight given before surgery, then 80 mg *3 for 48 hours after surgery.
  Interventions: Drug: Flucloxacillin and gentamicin

INTERVENTIONS:
Drug: Flucloxacillin and gentamicin — This intervention aimed to investigate the effectiveness of administering gentamicin in reducing the incidence of SSI.
  Arms: Gentamicin
Drug: Flucloxacillin and ceftriaxone — Control group
  Arms: Control

SUMMARY:
Surgical site infection (SSI) is a serious postoperative complication after cardiac surgery that have a negative impact on a patient's health and survival. This study aims to investigate the effectiveness of administering gentamicin in reducing the incidence of SSI with monitoring to the effective therapeutic level.

DETAILED DESCRIPTION:
Gentamicin is an aminoglycoside antibiotic that exhibits a wide range of antibacterial effects, mostly targeting Gram-negative bacteria, while its effectiveness against Gram-positive organisms is comparatively weaker. Gentamicin has significant efficacy against multidrug-resistant bacteria as well. Gentamicin is often used in conjunction with beta-lactam antibiotics to provide enhanced therapeutic efficacy via a synergistic effect, particularly in cases of Gram-positive and multidrug-resistant bacterial infections.

This study aims to evaluate the efficacy of administering gentamicin in combination with flucloxacillin as a pre-medication and for 48 hours after surgery in reducing the incidence of surgical site infections in patients undergoing cardiac surgeries, as compared to using a combination of ceftriaxone and flucloxacillin. Additionally, the study aimed to observes the therapeutic level of gentamicin required to achieve an effective concentration of the drug.

A prospective comparative study was conducted using an appropriate sample of 50 Iraqi patients undergone several types of cardiac surgeries.

A total of 50 patients (34 males and 16 females) between the ages of 18 and 75 were included in this study. These patients were admitted to the Surgical Department of the Iraqi Center for Heart Disease over a one-year period from January 2020 to January 2021. All patients underwent various types of cardiac surgery, such as coronary artery bypass graft (CABG), valve replacement, or device placement. The same surgical and anesthesia teams conducted the procedures.

A computerized randomization method was used to allocate patients into two groups in a randomized manner. Following the first interview, the patients were sequentially assigned numbers and then randomized into two groups via the online program Research Randomizer

ELIGIBILITY:
Inclusion Criteria:

* The research included individuals of both genders.
* Patients aged 18 and above.
* Patients had undergone any type of cardiac surgery.

Exclusion Criteria:

* Patients having a prior diagnosis of organ failure.
* Patients already on antibiotics.
* Patients with elevated baseline renal function test before operation.
* Patients with contraindications to any of the prescribed medications were excluded from this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
White blood cells | Up to 5 days post-surgery
  White blood cells count (WBCs per microliter).
Hemoglobin level | Up to 5 days post-surgery.
  Hemoglobin concentration (g/dl).
Erythrocyte sedimentation rate | Up to 5 days post-surgery.
  Erythrocyte sedimentation rate (millimeters per hour).
Body temperature | Up to 5 days post-surgery.
  Body temperature measurement (Degrees Celsius °C).

CONTACTS AND LOCATIONS:
Locations (1):
- Baghdad Medical City, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ackah JK, Neal L, Marshall NR, Panahi P, Lloyd C, Rogers LJ. Antimicrobial prophylaxis in adult cardiac surgery in the United Kingdom and Republic of Ireland. J Infect Prev. 2021 Mar;22(2):83-90. doi: 10.1177/1757177420971850. Epub 2020 Nov 24. PMID 33859725
- [Result] White RW, West R, Howard P, Sandoe J. Antimicrobial regime for cardiac surgery: the safety and effectiveness of short-course flucloxacillin (or teicoplanin) and gentamicin-based prophylaxis. J Card Surg. 2013 Sep;28(5):512-6. doi: 10.1111/jocs.12155. Epub 2013 Jul 9. PMID 23837413